CLINICAL TRIAL: NCT05064631
Title: Oral Bacterial Lysate to Prevent Persistent Wheeze in Infants After Severe Bronchiolitis; a Randomised Placebo-controlled Trial
Brief Title: Bacterial Lysate In Preventing Asthma
Acronym: BLIPA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Queensland University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 295882; 2021-000628-36 (EudraCT Number); NCT05710081 (obsolete NCT alias)
Record Dates: First submitted 2021-08-20; First posted 2021-10-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Tract Infections; Pediatric Respiratory Diseases; Wheezing
Keywords: Asthma in childhood; Bronchiolitis; Wheeze; Bacterial lysate
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Sounds; Bronchiolitis | interventions — Broncho-Vaxom

STUDY DESIGN:
Intervention Model Description: Children will be allocated into two arms (oral BV and placebo) in a 1:1 ratio. Randomisation will be stratified by site and parental asthma and the lists generated using random blocks of size 4 and 6.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parents or guardians will be blind to treatment allocation, as will the entire site study team involved in the management of the study, including the Chief Investigator (CI), PIs, sub-investigators, study nurses, and site coordinators. Trial Steering Committee (TSC) members will remain blind. The progress and safety of the study will be assessed by the Data Monitoring Committee (DMC). The DMC will therefore not be blinded. The main study trial manager (PCTU) and trial monitors will be blinded. The Sponsor's Joint Research Management Office (JRMO) including the JRMO monitor(s) will unblind themselves to specific patients in order to report SUSARs to the Medicines and Healthcare products Regulatory Agency (MHRA). The study pharmacist will be blinded, and the study pharmacy file will contain blinded documents, please see pharmacy manual. The treatment allocation list will be available from the PCTU or their designate (Sealed Envelope) on request should the need arise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active intervention (Experimental): Oral Broncho-Vaxom (3.5mg) administered daily for 10 days per month for 12-24 months
  Interventions: Drug: Bacterial Lysate
- Placebo control (Placebo Comparator): Matched placebo administered daily for 10 days per month for 12-24 months
  Interventions: Drug: Bacterial Lysate

INTERVENTIONS:
Drug: Bacterial Lysate — Bacterial lysate medicines are made from bacterial cells that are broken down and are intended to stimulate the immune system.
  Other Names: Broncho Vaxom

SUMMARY:
Bronchiolitis is a common viral infection of the small airways of infants and some affected infants will require hospital admission. Severe bronchiolitis is a marker for greatly increased risk of developing both preschool wheeze and subsequent school age asthma. Since epidemiological studies suggest that exposure to microbial products protects against preschool wheeze, lysates of bacteria may prevent the development of wheeze after bronchiolitis, with long-term beneficial consequences.

BLIPA is a phase 2b, randomised, double blind, placebo-controlled study, investigating the efficacy superiority of bacterial lysate (Broncho Vaxom) capsules over placebo, in reducing wheeze in infants after severe bronchiolitis. The primary end point of the study to establish whether there is superiority of oral Broncho-Vaxom over placebo in reducing the number of parent-reported wheeze episodes by 12 months post IMP/placebo initiation. The study aims to test bacterial lysate capsules (3.5mg over 12-24 months) for safety, efficacy, and to advance mechanistic understanding of its action.

DETAILED DESCRIPTION:
The BLIPA study aims to investigate the following research questions:

1. In children hospitalised with bronchiolitis, does Oral Broncho-Vaxom reduce incidence of parent-reported wheeze during 12 months post IMP initiation after a hospital admission for bronchiolitis.
2. Does oral BV reduces the risk of wheeze after bronchiolitis by modulating T cell and Dendritic cells (DC) maturation and altering the gut and airway microbiota. (mechanistic hypothesis)

The BLIPA study will combine the results of two multi-centre, randomised trials with similar but separate protocols: BLIPA-United Kingdom (UK), with recruitment in London, Southampton, Cheshire and Aberdeen and BLIPA-Australia, with recruitment in Brisbane, Gold Coast, Melbourne, Darwin and Sydney.

BLIPA-UK is funded in the UK by the NIHR (National Institute for Health and Care Research). BLIPA-Australia is funded in Australia by the International Clinical Trial Collaboration (ICTC). ICTC supports Australian researchers to conduct clinical trial research in collaboration with international researchers.

The total study duration is 74 months. The primary clinical objective is to recruit a population of eligible participants, to randomise them to oral Broncho Vaxom (3.5mg) or placebo, to be taken daily for 10 days a month over 12-24 months, follow up for 12-24 months and compare primary and secondary outcomes between trial arms. Parents or guardians of children, clinicians involved in their care and trial staff will be blinded to the treatment arm. Recruitment will be for 18 months and children's outcomes will be assessed for 24 months following initiation of Investigational Medicinal Product (IMP) or placebo.

Within six weeks of hospital discharge following admission for bronchiolitis, parents or guardians can consent to their child partaking in the study, baseline data is collected, the child is randomised, and the IMP or placebo is initiated (12 months' supply). From the point of treatment initiation, children are followed up for 12-24 months, the same length as the treatment period. There will be at least one scheduled face to face visit at 12 months to dispense a further year's supply of IMP or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Guardian able to provide written informed consent
* Within 6 weeks of discharge from hospital for bronchiolitis
* Child aged ≥2 weeks and ≤12 months at the time of consent to study
* A diagnosis of Bronchiolitis requiring a hospital admission (defined as more than 4 hours in hospital)
* Contactable for regular follow up by the research team

Exclusion Criteria:

* Any previous hospital attendance for bronchiolitis
* More than one episode of healthcare professional-diagnosed wheeze prior to index bronchiolitis episode
* Premature gestational age less than 37 weeks
* Any severe chronic condition such as cystic fibrosis, sickle cell disease, severe developmental delay, immunodeficiency, or anything that has a significant impact on the respiratory tract (such as need for non-invasive ventilation) or increases vulnerability to respiratory tract infections.
* History of clinically significant neonatal disease (e.g. neonatal pneumonia, congenital lung abnormality, neonatal chronic lung disease)
* Genetic conditions that affect the immune system (e.g. Down's syndrome/Trisomy 21)
* Current regular oral montelukast or inhaled corticosteroid therapy or inhaled salbutamol therapy
* Current regular treatment with immunomodulatory drugs (e.g oral steroids)
* Known allergy or previous intolerance to study medication.
* Currently enrolled to another Randomised Clinical Trial. (Unless prior approval is given by Principal Investigator)
* Sibling of a BLIPA participant (of the same household or family)

Ages: 2 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of a wheeze episodes by 12 months | 12 months
  To establish whether there is superiority of oral Broncho-Vaxom over placebo in the reduction of parent reported wheeze episodes by 12 months post IMP/placebo initiation

SECONDARY OUTCOMES:
To establish whether there is a difference between treatment with Broncho-Vaxom or placebo in healthcare professional confirmed wheeze episodes by 12 months post IMP initiation. | 12 months
  Wheeze confirmed via one of the following:
  1. Prescription for more than one salbutamol inhaler coded in primary care record between 0-12 months post IMP/placebo initiation.
  2. Active wheeze code in primary care records between 0-12 months post IMP/placebo initiation.
  3. Asthma diagnosis code in primary care records between 0-12 months post IMP/placebo initiation.
Occurrence of hospital admissions for wheeze-related illness by 12 months. | 12 months
  Occurrence of hospital admissions for wheeze-related illness by 12 months.
Occurrence of unscheduled medical attendance for wheeze-related illness by 12 months | 12 months
  Occurrence of unscheduled medical attendance for wheeze-related illness (rate[episodes per child/month] and yes/no).
Presence of wheeze diagnosis by 12 months | 12 months
  Presence of wheeze diagnosis by 12 months
Time to first wheeze episode by 12 months | 0-12 months
  Time to first wheeze episode by 12 months
Duration of wheeze by 12 months | 12 months
  Duration of wheeze by 12 months
Development of eczema by 12 months | 12 months
  Development of eczema by 12 months confirmed by parent report at study follow ups (parent reported outcome)
Development of Dr-diagnosed food allergy by 12 months | 12 months
  Development of Dr-diagnosed food allergy by 12 months
Occurrence of all-cause acute respiratory infection by 12 months | 12 months
  Occurrence of all-cause acute respiratory infection by 12 months
Hospital admissions for respiratory related illness (rate[episodes per child-month] and yes/no) by 12 months | 12 months
  Hospital admissions for respiratory related illness (rate[episodes per child-month] and yes/no) by 12 months
Quality of life confirmed by Warwick Child Health and Morbidity by 12 months | 12 months
  Quality of life confirmed by Warwick Child Health and Morbidity by 12 months
Number of courses of oral corticosteroids for wheeze by 12 months | 12 months
  Number of courses of oral corticosteroids for wheeze by 12 months
Incidence of adverse events (AEs) for the treatment group by 12 months | 12 months
  Number of AEs by 12 months
Incidence of serious adverse events (SAEs) for the treatment group by 12 months | 12 months
  Number of SAEs by 12 months
Incidence of Suspected unexpected serious adverse reactions (SUSARs) for the treatment group by 12 months | 12 months
  Number of SUSARs by 12 months
Incidence of adverse events (AEs) for the treatment group between 0-24 months | 0-24 months
  Number of AEs across 0-24 months
Incidence of serious adverse events (SAEs) for the treatment group between 0-24 months | 0-24 months
  Number of SAEs across 0-24 months
Incidence of Suspected unexpected serious adverse reactions (SUSARs) for the treatment group between 0-24 months | 0-24 months
  Number of SUSARs across 0-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grigg, Prof. Dr, Study Chair — Queen Mary University of London
Locations (3):
- United Kingdom (3):
  - Royal London Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No